CLINICAL TRIAL: NCT07135193
Title: Evaluation of the Protective Effects of Cordyceps Cicadae on Visual Function and Anti-Fatigue Performance in Esports Athletes: A Prospective Trial
Brief Title: Evaluation of the Protective Effects of Cordyceps Cicadae on Visual Function and Anti-Fatigue Performance in Esports Athletes
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Principal Investigator, Hui Wen Lin, Ph.D, China Medical University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: CS1-25024
Record Dates: First submitted 2025-08-11; First posted 2025-08-21 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Visual Acuity; Accommodation; Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Arm (Experimental): Cordyceps cicadae 500mg
  Interventions: Dietary Supplement: Cordyceps cicadae
- Placebo Comparator Arm (Placebo Comparator): Placebo
  Interventions: Dietary Supplement: Blank control

INTERVENTIONS:
Dietary Supplement: Cordyceps cicadae — Cordyceps cicadae 500mg
  Arms: Experimental Arm
Dietary Supplement: Blank control — Blank control
  Arms: Placebo Comparator Arm

SUMMARY:
The objective of this study is to evaluate, through a clinical human consumption trial, the effects of taking two capsules (each containing 250 mg of Cordyceps cicadae mycelium, for a total intake of 500 mg per dose) of Grape King Cordyceps cicadae mycelium on visual function and anti-fatigue performance in esports athletes.

DETAILED DESCRIPTION:
This study aims to enroll 12 participants (aged 20-30 years), who are esports players, through oral announcements for recruitment. The anticipated source of participants will be students from the Department of Multimedia Game Development and Applications, Hungkuang University of Science and Technology, second-year and above.

On the day prior to the trial, participants will undergo a baseline ophthalmic examination (serving as the control values). Following the baseline assessment, participants will undergo ophthalmic examinations after 1 hour and 2 hours of esports training, respectively, resulting in a total of three measurements. All data will be recorded in the case report form (CRF).

On the day of the trial, participants will first undergo an ophthalmic examination. After completion, all 12 participants will be randomly allocated into groups using the QuickCalcs randomization tool (GraphPad Software, https://www.graphpad.com/quickcalcs/randomize1/). Based on the random allocation, capsule packages labeled with codes 001 to 012 will be prepared, containing either the investigational product or placebo. Each package will be distributed to the corresponding participant. Of the 12 participants, 3 will be assigned to the placebo group, and 9 will be assigned to the Cordyceps cicadae mycelium group.

Participants will undergo ophthalmic examinations at 1 hour and 2 hours post-administration, and the results will be recorded in the CRF.

The investigational product will be in capsule form, containing Cordyceps cicadae mycelium (250 mg per capsule) and excipients, with no other additives. The placebo will have the same excipients and capsule composition, except without the mycelium. Each participant will take a single oral dose on the test day (2 capsules). All investigational products and placebos will be provided by Grape King Bio Ltd.

ELIGIBILITY:
Inclusion Criteria:

* People with myopia less than 700 degrees
* Willing to participate in this study and sign the consent form

Exclusion Criteria:

* (1) Those who have recently consumed related eye care products
* (2) Those who have had eye infections or surgery in the past three months
* (3) Those who have been diagnosed with eye diseases by an ophthalmologist (such as glaucoma, cataracts, macular degeneration, diabetic retinopathy, etc., or have undergone eye surgery such as cataract surgery, retinal laser surgery, myopia laser surgery, etc., which will be excluded before accepting the case)
* (4) Those who are allergic to cicada fungus

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2025-08-12 (Actual); Primary Completion 2025-08-13 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Tear break-up time | 3 hours
  Tear film break-up time (TBUT) on the corneal surface will be recorded in seconds using corneal topography.
Eye fatigue questionnaire | 3 hours
  The Ocular Surface Disease Index (OSDI) was used to assess visual fatigue. The subjects were asked to fill in the questionnaire before and after taking the medicine, and the scores were calculated. Symptoms include eyestrain, discomfort, burning, irritation, pain, soreness, eye pain, double vision, photophobia, blurriness, itching, tearing, dryness, and foreign body sensation
Accommodative Facility | 3 hours
  Use +/- 0.50D flip mirror and special optometry cards to test the number of optometry cards that the patient can read within one minute and record the number of flip cycles.
Visual acuity measurement | 3 hours
  Examinations include (a) distance visual acuity (DVA) and (b) near visual acuity (NVA), recorded using the Snellen chart.
Intraocular Pressure | 3 hours
  The intraocular pressure (IOP) of the subjects was measured by non-contact intraocular pressure measurement in mmHg.
Tear meniscus height (TMH) | 3 hours
  Tear meniscus height (TMH) will be evaluated using slit-lamp biomicroscopy and recorded in millimeters.
Meibomian gland observation | 3 hours
  The meibomian glands will be evaluated using corneal topography to document their morphology, quantity, and size.

CONTACTS AND LOCATIONS:
Overall Officials: Hui-Wen Lin, Ph.D, Principal Investigator — Chung Shang medical university
Locations (1):
- Chung Shan Medical University Hui-Wen Lin lab, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No
This experiment involves patents and intellectual property rights